CLINICAL TRIAL: NCT02004509
Title: SILENT - Subclinical AtrIal FibrilLation and StrokE PreveNtion Trial
Brief Title: Subclinical AtrIal FibrilLation and StrokE PreveNtion Trial
Acronym: SILENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Martino Martinelli Filho, Prof., MD, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILENT
Record Dates: First submitted 2013-09-24; First posted 2013-12-09 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; stroke; pacemaker; anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anticoagulant (Active Comparator): Prescription of oral anticoagulation for patients with silent AF (detected by the pacemaker).
  Interventions: Drug: Anticoagulant
- Control (No Intervention): Patients with silent FA detected only by the pacemaker will no receive oral anticoagulation.

INTERVENTIONS:
Drug: Anticoagulant — Anticoagulant treatment will be started in case of subclinical atrial fibrillation (>5,5 hours per day) be diagnosed by cardiac implantable electronic device at intervention group, or clinical atrial fibrillation in both groups.
  Other Names: Oral Anticoagulant
  Arms: anticoagulant

SUMMARY:
Introduction: Patients with atrial fibrillation (AF) have a substantial risk of stroke and systemic embolism. Subclinical AF is often suspected to be the cause of stroke in these patients. The detection of asymptomatic AF episodes is a challenge and the real rate of occurrence of these episodes remains unknown. The rate of stroke is high among patients who have received a pacemaker and this device can detect subclinical episodes of rapid atrial rate, which correlate with electrocardiographically documented AF. The net benefit of anticoagulant treatment is well established in patients with clinical AF but data about anticoagulation in subclinical AF setting is unknown. The aim of this study is to assess the impact of anticoagulant therapy on subclinical AF, directed by cardiac implantable electronic device (CIED) intensive monitoring, on the incidence of stroke and systemic embolism and correlate the AF episodes detected by CIED with thromboembolic events. Methods: This is a prospective, randomized, unicentric, parallel clinical study in patients with atrioventricular pacemaker, defibrillator, or cardiac resynchronization therapy devices in sinus rhythm and CHADS2 score (an index of the risk of stroke in patients with atrial fibrillation, range from 0 to 6) ≥ 2 . Patients will be randomized to the intervention group - intensive monitoring arm (Group I) or control group - routine schedule arm (Group II) in a 1:1 ratio. Time to inclusion will be 24 months and all patients will be followed up for a period of 36 months. Group I, patients will be submitted to device data collection every 2 months, while in Group II, patients will be managed conventionally. Patients from Group I with episodes of subclinical AF will receive anticoagulant therapy, as well as patients with clinical AF of both arms. Device data from Group II patients will not be analyzed until they achieve the primary endpoint. Primary endpoint: stroke or systemic embolism. Secondary endpoints: subclinical AF rate, total mortality, cardiovascular mortality, myocardial infarction, cardiovascular hospitalization, and bleeding rates. Expected outcome: It is expected that anticoagulation therapy of subclinical AF directed by CIED intensive monitoring will reduce the incidence of stroke and systemic embolism comparing to patients with non-diagnosed subclinical AF.

DETAILED DESCRIPTION:
Patients with atrial fibrillation (AF) have a substantial risk of stroke and systemic embolism. Subclinical AF is often suspected to be the cause of stroke in these patients. The detection of asymptomatic AF episodes is a challenge and the real rate of occurrence of these episodes remains unknown. The rate of stroke is high among patients who have received a pacemaker and this device can detect subclinical episodes of rapid atrial rate, which correlate with electrocardiographically documented AF. The net benefit of anticoagulant treatment is well established in patients with clinical AF but data about anticoagulation for subclinical AF settings is unknown. The aim of this study is to assess the impact of anticoagulant therapy on subclinical AF, directed by cardiac implantable electronic device (CIED) intensive monitoring, on the incidence of stroke and systemic embolism and correlate the AF episodes detected by CIED with thromboembolic events. Methods: This is a prospective, randomized, unicentric, parallel clinical study in patients with an atrioventricular pacemaker, defibrillator, or cardiac resynchronization therapy devices in sinus rhythm and CHADS2 score (an index of the risk of stroke in patients with atrial fibrillation, range from 0 to 6) ≥ 2 . Patients will be randomized to the intervention group - intensive monitoring arm (Group I) or control group - routine schedule arm (Group II) in a 1:1 ratio. Time to inclusion will be 24 months and all patients will be followed up for a period of 36 months. Group I, patients will be submitted to device data collection every 2 months, while in Group II, patients will be managed conventionally. Patients from Group I with episodes of subclinical AF will receive anticoagulant therapy, as well as patients with clinical AF of both arms. Device data from Group II patients will not be analyzed until they achieve the primary endpoint. Primary endpoint: stroke or systemic embolism. Secondary endpoints: subclinical AF rate, total mortality, cardiovascular mortality, myocardial infarction, cardiovascular hospitalization, and bleeding rates. Expected outcome: It is expected that anticoagulation therapy of subclinical AF directed by CIED intensive monitoring will reduce the incidence of stroke and systemic embolism comparing to patients with non-diagnosed subclinical AF.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* CHADS2 score >=2
* Sinus rhythm
* Cardiac Implantable Electronic Device

Exclusion Criteria:

* Atrial fibrillation
* Severe heart valve disease
* Anticoagulation therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2054 (Estimated)
Dates: Start 2015-02-06 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | 36 months
  Occurrence of stroke
Systemic embolism | 36 months
  Occurrence of systemic embolism

SECONDARY OUTCOMES:
Subclinical AF rate | 36 months
  Rate subclinical AF documentation by pacemaker
Total mortality | 36 months
  All cause mortality
Cardiovascular mortality | 36 months
  Adjudicated cardiovascular mortality
Myocardial infarction | 36 months
  Occurrence of myocardial infarction
Cardiovascular hospitalization | 36 months
  Adjudicated cardiovascular hospitalization
Bleeding rates | 36 months
  Occurrence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Sergio F Siqueira, Eng, Study Director — Biomedical Eng
Locations (1):
- Martino Martinelli Filho, São Paulo, São Paulo, Brazil